CLINICAL TRIAL: NCT00632762
Title: Evaluation of the Long-term Effects of Amantadine in Parkinsonian's Suffering From Dyskinesia Induced by Levodopa: Study Randomised Double-blind, Placebo - Cessation of a Chronic Prescription. STUDY AMANDYSK.
Brief Title: Long-Term Effects of Amantadine in Parkinsonian (AMANDYSK)
Acronym: AMANDYSK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Marie-Elise LLAU, UH TOULOUSE
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06 008 01
Record Dates: First submitted 2008-02-20; First posted 2008-03-11 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Parkinson's Disease
Keywords: Amantadine benefit; Dyskinesia; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Amantadine MANTADIX
  Interventions: Drug: mantadix
- 2 (Placebo Comparator): placebo
  Interventions: Drug: mantadix

INTERVENTIONS:
Drug: mantadix — dose greater or equal to 200 mg/day and progressively increasing doses (100mg every 3 days until the pre-study dose is reached).

SUMMARY:
This is a French national trial, conducted using a double-blind, placebo-controlled, randomised design involving 7 centers and 80 patients of both sexes.

The primary objective of the trial is to evaluate the effects of the interruption of a long term treatment (ex. Greater than 6 months) with Amantadine (prescribed as an antidyskinetic) in patients suffering from Parkinson disease being treated with Levodopa and suffering from mid dose dyskinesias.

Secondary objectives of the trial are the evaluation of the other effects of withdrawal of Amantadine on the same group of patients: motor fluctuations, vigilance, apathy, fatigue, certain cognitive aspects, the disappearance or development of undesirable side effects and quality of life.

DETAILED DESCRIPTION:
The trial will involve the participation of the patients for a period of 3 months each. The two groups of patients to be studied are:

* a group who will continue their treatment with Amantadine with no modification to dosage;
* a group who will have their dosage of Amantadine progressively replaced over several days with a placebo (with the aim of avoiding a "brutal" withdrawal which has been associated with symptoms of hyperthermia in rare cases in the literature).

The trial visits are scheduled as such:

* weekly visits for the first 4 weeks, with a telephone call between each visit to assure that the withdrawal from Amantadine causes any problems.
* every 2 weeks from week 4 until week 8, with weekly telephone calls in between these visits.
* a telephone call in the 10th week followed by an end of study visit in week 12. In the event of an early withdrawal from the trial, and assuming that the patient gives their consent, a complete end of study visit will be performed prior to recommencing open label treatment with Amantadine in progressively increasing doses (100mg every 3 days until the pre-study dose is reached).

ELIGIBILITY:
Inclusion Criteria:

* Female or Male Patients with Idiopathic Parkinson's disease
* Presenting peak dose dyskinesias under levodopa therapy
* Patient receiving Amantadine for dyskinesia at a dose greater or equal to 200 mg/day (minimum dose at which one can observe anti dyskinetic effects) for at least 6 months.
* Patients between 30 and 80 years of age
* Patients having reported a subjective amelioration in their dyskinesias under Amantadine (at the beginning of their treatment with same)
* Patient with a Mini- Mental State Exam score > 24
* Patient not presenting a cognitive problem that could impair the comprehension of the patient and their participation in the protocol (patient diaries)
* Receiving an anti-parkinsonian treatment at a stable dose for at least 2 months with the expectation that the treatment will remain unchanged throughout the course of the patients participation in the trial.
* Signed informed consent obtained
* Patient eligible for social security (specific requirement under french law)

Exclusion Criteria:

* Atypical parkinsonian syndrome (progressive supranuclear palsy, multi-system atrophy, etc)

  * Patient with parkinsonian syndrome secondary to medication
  * Patients presenting with dyskinesias whose severity allow an insufficient margin for observing any aggravation which follows a potential withdrawal of treatment (UPDRS 32+33 >6)
  * Patients receiving treatment with Apokinon© injector pens (unless that treatment enters into a therapeutic schema at fixed hours)
  * Patient presenting with dementia or an evolving dopaminergic psychosis
  * Patient receiving neuroleptics or anticholinesterases
  * Patients having received functional surgery for their Parkinsons' Disease
  * Patients pregnant or at risk of same
  * Patients who are: wards of the state requirement under french law).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the variation in the sum of the items 32 and 33 (duration and severity of dyskinesias - maximum score = 8) evaluated using Part IV of the UPDRS scale | 3 months

SECONDARY OUTCOMES:
The number of patient "responders" | 3 months
The number of premature withdrawals from the trial for reason of an aggravation of dyskinesias | 3 months
The AIMS scale | 3 months
The Clinical Global Impression Severity Scale | 3 months
Other "exploratory" secondary efficacy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, MD, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - Hôpital d'Aix en Provence, Aix-en-Provence
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Timone, Marseille
  - Hôpital Haut-Lévêque, Nantes
  - CHU Pitié-Salpêtrière, Paris

REFERENCES:
- [Background] Alves G, Wentzel-Larsen T, Larsen JP. Is fatigue an independent and persistent symptom in patients with Parkinson disease? Neurology. 2004 Nov 23;63(10):1908-11. doi: 10.1212/01.wnl.0000144277.06917.cc. PMID 15557510
- [Background] Bibbiani F, Oh JD, Kielaite A, Collins MA, Smith C, Chase TN. Combined blockade of AMPA and NMDA glutamate receptors reduces levodopa-induced motor complications in animal models of PD. Exp Neurol. 2005 Dec;196(2):422-9. doi: 10.1016/j.expneurol.2005.08.017. Epub 2005 Oct 3. PMID 16203001
- [Background] Chapuis S, Ouchchane L, Metz O, Gerbaud L, Durif F. Impact of the motor complications of Parkinson's disease on the quality of life. Mov Disord. 2005 Feb;20(2):224-30. doi: 10.1002/mds.20279. PMID 15384126